| Document Type: | Statistical Analysis Plan |
|---|---|
| Official Title: | A Phase 2, Open-Label Study of HTX-011 in a Multimodal Analgesic<br>Regimen for Decreased Opioid Use Following Unilateral Open Inguinal<br>Herniorrhaphy |
| NCT Number: | NCT03695367 |
| Document Date: | 18-Oct-2018 |

Clinical Study Report: HTX-011-215 Phase 2 Herniorrhaphy Study for Opioid Elimination

#### **Documentation of Statistical Methods** 16.1.9.

Statistical Analysis Plan Version 1.0 dated 18 October 2018

Confidential Page 1 of 28

## STATISTICAL ANALYSIS PLAN

## HTX-011-215

A Phase 2, Open-Label Study of HTX-011 in a Multimodal Analgesic Regimen for Decreased Opioid Use Following Unilateral Open Inguinal Herniorrhaphy

Prepared by:

Heron Therapeutics, Inc. 4242 Campus Point Court, Suite 200 San Diego, CA 92121 USA

Version 1: 18 October 2018

Upon review of this document, the undersigned approves the statistical analysis plan. The analysis methods are acceptable, and the table, listing, and figure shell production can begin.

| Approved by: | Date: | |
|---|---|---|
| | Vice President, Biometrics<br>Heron Therapeutics, Inc. | |
| Approved by: | | Date: |
| | Vice President, Clinical Research<br>Heron Therapeutics, Inc. | |

#### **Confidentiality Statement**

This document contains confidential information of Heron Therapeutics, Inc.

Do not copy or distribute without written permission of the Sponsor.

Any authorized use, reproduction, publication, or dissemination is strictly prohibited.

# TABLE OF CONTENTS

| 1. | ADMINISTRATIVE STRUCTURE | 7 |
|--------|--------------------------------------------------------|----|
| 1.1. | Sponsor and Oversight | 7 |
| 1.2. | Data Quality Assurance | 7 |
| 2. | INTRODUCTION | 7 |
| 3. | OBJECTIVES | 7 |
| 4. | INVESTIGATIONAL PLAN | 8 |
| 4.1. | Overall Study Design and Plan | 8 |
| 4.2. | Assessments | 8 |
| 4.3. | Endpoints | 9 |
| 4.3.1. | Efficacy Endpoints | 9 |
| 4.3.2. | Safety Endpoints | 9 |
| 5. | GENERAL STATISTICAL CONSIDERATIONS | 10 |
| 5.1. | Sample Size | 10 |
| 5.2. | Randomization, Stratification, and Blinding | 10 |
| 5.3. | Analysis Populations | 11 |
| 5.3.1. | Safety Population | 11 |
| 5.4. | Other Important Considerations | 11 |
| 5.4.1. | Definition of Baseline | 11 |
| 5.4.2. | Calculation of Change and Percent Change from Baseline | 11 |
| 5.4.3. | Study Day Calculation for Reporting Purposes | 11 |
| 5.4.4. | Start date/time of Study Drug Administration (Time 0) | 11 |
| 5.4.5. | 72-Hour Postoperative Observation Period | 11 |
| 5.4.6. | Visit Windows | 12 |
| 5.4.7. | Handling of Missing and Partial Data | 12 |
| 6. | SUBJECT DISPOSITION | 12 |
| 7. | DEMOGRAPHICS, CHARACTERISTICS, AND MEDICAL HISTORY | 13 |
| 7.1. | Demographics and Baseline Characteristics | 13 |
| 7.2. | Medical History | 13 |
| 7.3. | Protocol Deviations | 13 |
| 8. | TREATMENTS AND MEDICATIONS | 13 |
| 8.1. | Prior and Concomitant Medications | 13 |

| 8.2. | Surgery Procedure | 14 |
|---|---|---|
| 8.3. | Study Drug | 14 |
| 9. | EFFICACY ANALYSIS | 14 |
| 9.1. | Primary Efficacy Endpoint | 14 |
| 9.1.1. | Primary Analysis | 14 |
| 9.2. | Secondary Efficacy Endpoints | 15 |
| 10. | SAFETY ANALYSIS | 17 |
| 10.1. | Adverse Events | 17 |
| 10.1.1. | Incidence of Treatment Emergent Adverse Events | 18 |
| 10.1.2. | Relationship of Adverse Events to Investigational Drug | 18 |
| 10.1.3. | Severity of Adverse Event | 19 |
| 10.1.4. | Serious Adverse Events | 19 |
| 10.1.5. | Adverse Events Leading to Study Withdrawal | 19 |
| 10.1.6. | Opioid-related Adverse Events | 19 |
| 10.1.7. | Local Inflammatory Adverse Events | 20 |
| 10.1.8. | Potential Local Anesthetic Systemic Toxicity (LAST) related Adverse Events | 20 |
| 10.1.9. | Death | 20 |
| 10.2. | Clinical Laboratory Evaluations | 21 |
| 10.3. | Hematology | 21 |
| 10.3.1. | Blood Chemistry | 21 |
| 10.3.2. | Urine Pregnancy Test and Urine Drug Screen | 22 |
| 10.4. | Vital Sign Measurements | 22 |
| 10.5. | Electrocardiogram | 23 |
| 10.6. | Physical Examination | 23 |
| 10.7. | Wound Healing Assessment | 23 |
| 11. | INTERIM ANALYSIS | 24 |
| 11.1. | Interim Analysis | 24 |
| 11.2. | Data Safety Monitoring Board | 24 |
| 12. | REFERENCES | 24 |
| APPENI | DIX 1. IMPUTATION OF PARTIAL AND MISSING DATES | 25 |
| APPENI | DIX 2. DOCUMENT REVISION HISTORY | 26 |

# LIST OF TABLES

| Table 1. | Analgesic Windows and IV Morphine Milligram Equivalents for Opioid | |
|---|---|---|
| | Rescue Medications in Preferred Terms | 16 |
| Table 2. | Local Inflammatory Adverse Events by Preferred Term | 20 |
| Table 3. | Potential LAST-Related Adverse Events by Preferred Term | 20 |
| Table 4. | Clinically Relevant Vital Signs Abnormalities | 23 |

# List of Abbreviations

| Abbreviation | Term |
|--------------|---------------------------------------------------|
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| ATC | Anatomic Therapeutic Classification |
| AUC | Area under the curve |
| bpm | Beats per minute |
| BMI | Body mass index |
| BUN | Blood urea nitrogen |
| CRO | Contract research organization |
| CSR | Clinical Study Report |
| DBP | Diastolic blood pressure |
| DM | Data management |
| DSMB | Data Safety Monitoring Board |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| eDISH | Evaluation of drug-induced serious hepatotoxicity |
| GGT | Gamma-glutamyltransferase |
| IV | Intravenous(ly) |
| LAST | Local Anesthetic Systemic Toxicity |
| LOCF | Last observation carried forward |
| MCV | Mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MME | Morphine milligram equivalent |
| NRS | Numeric Rating Scale |
| NRS-R | Numeric Rating Scale at rest |
| NSAID | Nonsteroidal anti-inflammatory drug |
| ORAE | Opioid-related adverse event |
| PT | Preferred term |
| RBC | Red blood cell |
| SAE | Serious adverse event |

| Abbreviation | Term |
|--------------|----------------------------------------------------|
| SAP | Statistical Analysis Plan |
| SBP | Systolic blood pressure |
| SD | Standard deviation |
| SDA | Study drug administration |
| SDTM | Study Data Tabulation Model |
| SDTMIG | Study Data Tabulation Model Implementation Guide |
| SE | Standard error |
| SOC | System Organ Class |
| TEAE | Treatment-emergent adverse event |
| ULN | Upper limit of normal |
| WBC | White blood cell |
| WHODDE | World Health Organization Drug Dictionary Enhanced |
| wWOCF | Windowed worst observation carried forward |

#### 1. ADMINISTRATIVE STRUCTURE

## 1.1. Sponsor and Oversight

This study is being conducted under the sponsorship of Heron Therapeutics, Inc. (Heron).

## 1.2. Data Quality Assurance

The DM and Biostatistics departments at the contract research organizations (CROs) will collaborate internally and with the Sponsor to ensure that the data collected and analyzed for this study are of the highest quality possible and meet the data standards set for the study. This will be accomplished in part through programmed edit checks which will be reviewed by the data managers, statisticians, programmers, and other team members on an ongoing basis to evaluate whether any checks need to be added or any existing checks need to be modified. In addition, periodic reviews of listings of accumulating data, assessment of data query trends, and resulting retraining of study site personnel will be performed to further ensure data quality.

#### 2. INTRODUCTION

This statistical analysis plan (SAP) presents a detailed plan of the statistical methods to be used for the reporting of efficacy and safety data collected in this study.

This SAP was prepared prior to data analysis to provide full details of analyses to be presented in the clinical study report (CSR), including a detailed elaboration of the statistical analysis methods presented in the protocol. Revisions can be made to this SAP while the study is ongoing; however, it must be finalized prior to database lock. Any deviations from the analysis plan provided in the SAP will be fully documented in the final CSR.

This SAP should be read in conjunction with the study protocol and the electronic Case Report Forms (eCRFs).

#### 3. OBJECTIVES

The primary objective of the study is as follows:

To assess the proportion of subjects who are opioid-free after receiving HTX-011
as part of a multimodal analgesic regimen during the first 72 hours following
unilateral open inguinal herniorrhaphy with mesh.

The secondary objectives are as follows:

- To assess the total opioid use following HTX-011 as part of a multimodal analgesic regimen during the first 72 hours following surgery in this study population.
- To assess the proportion of subjects who are opioid-free after receiving HTX-011 as part of a multimodal analgesic regimen during the first 72 hours that remain opioid-free through Day 10 and Day 28.
- To assess the relationship between opioid use and severe pain.

#### 4. INVESTIGATIONAL PLAN

## 4.1. Overall Study Design and Plan

This is a Phase 2 open-label study in subjects undergoing unilateral open inguinal herniorrhaphy in up to 3 cohorts. See the study protocol, Section 3.1.3 for a description of the inpatient scheduled analgesic regimen and the discharge/postoperative analgesic regimen for all cohorts.

#### Cohort 1

Approximately 30 subjects will be enrolled and dosed in one treatment group:

• HTX-011 300 mg/9 mg (bupivacaine/meloxicam doses), 10.3 mL, via instillation into the surgical site.

#### **Optional Cohort 2**

At the Sponsor's discretion upon completion of Cohort 1, Optional Cohort 2 may be initiated. If conducted, Optional Cohort 2 will be composed of approximately 30 subjects. Optional Cohort 2 would consist of the same required preoperative, intraoperative, and scheduled pain medication regimen as in Cohort 1 would be required with the intra-operative addition prior to wound closure of 1 dose of IV ketorolac as follows:

- For subjects aged ≥65 years, Serum Creatinine >1.5, and/or weight <50 kg: 15 mg.
- For subjects aged <65 years and/or weight ≥50 kg: 30 mg.

#### **Optional Cohort 3**

At the Sponsor's discretion upon completion of Optional Cohort 2, Optional Cohort 3 may be initiated. If conducted, Optional Cohort 3 will be composed of approximately 30 subjects. The specific multimodal analgesic regimen in Optional Cohort 3 will be determined by the Sponsor and included in a protocol amendment.

#### 4.2. Assessments

Efficacy assessments will include the following:

• Pain intensity scores using the NRS at rest (NRS-R).

• Use of opioid rescue medication.

Safety assessments will include the following:

- Adverse event (AE) recording.
- Concomitant medication recording.
- Clinical safety laboratory tests (hematology and serum chemistry).
- 12-lead electrocardiogram (ECG).
- Physical examination.
- Wound healing assessment.
- Vital signs collections.

## 4.3. Endpoints

### 4.3.1. Efficacy Endpoints

The primary efficacy endpoint is the following:

• Proportion of subjects receiving no opioid rescue from 0-72 hours.

The secondary efficacy endpoints are the following:

- Total postoperative opioid consumption (in IV morphine milligram equivalents [IV MME]) through 72 hours.
- Proportion of subjects receiving no opioid rescue over the following time intervals: 0-24 hours, 24-48 hours, 0-48 hours, 24-72 hours, 48-72 hours.
- Proportion of subjects receiving no opioid rescue from 0-72 hours who receive no opioid rescue through Day 10, and through Day 28.
- Proportion of subjects in severe pain (NRS-R  $\geq$ 7) at any point in the first 72 hours postoperatively.

#### 4.3.2. Safety Endpoints

The safety endpoints are the following:

- Incidence of treatment-emergent AEs (TEAEs), serious TEAEs (SAEs), and opioid-related AEs (ORAEs) through Day 28.
- Change from baseline in clinical laboratory results.
- Change from baseline in ECG data.
- Change from baseline in vital signs.
- Wound healing assessment at 72 hours and on Day 10 and 28.

#### 5. GENERAL STATISTICAL CONSIDERATIONS

No statistical hypothesis testing will be performed. Continuous data will be presented using descriptive statistics: number of subjects (n), mean, standard deviation (SD), median, minimum and maximum. Descriptive statistics on efficacy measures will also include the standard error (SE). Categorical data will be summarized by the number and percent of subjects. Data will be displayed in all listings sorted by cohort, subject number and visit/study day. When count data are presented, the percent will be suppressed when the count is zero in order to draw attention to the non-zero counts. A row denoted "Missing" will be included in count tabulations where necessary to account for dropouts and missing values. The denominator for all percentages will be the number of subjects in that treatment group within the population of interest, unless otherwise stated. Non-zero percentages will be rounded to 1 decimal place, except 100% will be displayed without any decimal places. Additional rounding rules are as follows:

- If the original value has 0 decimal places: mean, median, and CI will have 1 decimal place and SD and SE will have 2 decimal places.
- If the original value has 1 decimal place: mean, median, and CI will have 2 decimal places and SD and SE will have 3 decimal places.
- If the original value has 2 or more decimal places: mean, median, CI, SD, and SE will all have 3 decimal places.

Minimum and maximum will always have the same decimal places as the original measure, up to a maximum of 3 decimal places. The above rounding rules will not be applied to original measures displayed in listings.

Values that are collected with "<" or ">" signs will be analyzed as the numerical value without the sign in tables and figures. In listings, these data will be reported as collected with the sign.

All efficacy and safety data will be collected electronically. Datasets will be created using the Study Data Tabulation Model (SDTM) v. 1.4 or higher, conforming to the SDTM Implementation Guide (SDTMIG) v. 3.2 or higher. Datasets, tables, listings, and figures will be programmed using SAS® v. 9.4 or higher. All efficacy and safety data will be listed via the SDTM datasets and selected efficacy and safety data will be listed via programmed listings.

## 5.1. Sample Size

The sample size in this study was selected empirically without a formal statistical assumption.

## 5.2. Randomization, Stratification, and Blinding

This is an open-label study.

## 5.3. Analysis Populations

#### **5.3.1.** Safety Population

The Safety Population will consist of all subjects who receive study drug. This population will be used for all summaries of efficacy and safety data.

## **5.4.** Other Important Considerations

#### **5.4.1.** Definition of Baseline

Baseline data are defined as the last observed measurement collected, whether scheduled or unscheduled, prior to the start of study drug administration.

#### 5.4.2. Calculation of Change and Percent Change from Baseline

Change from Baseline to any timepoint t (C<sub>t</sub>) is calculated as follows:

$$C_t = M_t - M_B$$
, where:

- M<sub>t</sub> is the measurement of interest at timepoint t.
- M<sub>B</sub> is the measurement of interest at Baseline.

Percent change from Baseline to any timepoint  $(P_t)$  is calculated as follows:

$$P_t = 100*(C_t/M_B)$$

#### 5.4.3. Study Day Calculation for Reporting Purposes

The following convention will be used to calculate study day for reporting purposes:

- The study day of study drug administration is Study Day 1.
- For measurements that are *on or after* the date of study drug administration:
  - Study Day = date of measurement date of study drug administration + 1.
- For measurements that are *prior* to the date of study drug administration:
  - Study Day = date of measurement date of study drug administration.

For all subjects, the day of study drug administration should be the same day as the day of the surgical procedure.

#### 5.4.4. Start date/time of Study Drug Administration (Time 0)

The start date/time of study drug administration is defined as the date and time of the start of HTX-011 instillation. The start date/time of study drug administration will be Time 0 for all efficacy and safety assessments.

#### 5.4.5. 72-Hour Postoperative Observation Period

The 72-hour postoperative observation period will be defined as the period of time from the start date/time of study drug administration to the date/time of NRS-R pain intensity score assessment at the nominal 72-hour postoperative timepoint.

Subjects who have a reported NRS-R pain intensity score at the nominal 72-hour postoperative timepoint will be considered as completing the 72-hour postoperative observation period.

#### 5.4.6. Visit Windows

Due to the short duration of the study and the primary efficacy analyses occurring during the 72-hour postoperative period of subject hospitalization, no programmatically calculated visit windows are defined for this study.

#### 5.4.7. Handling of Missing and Partial Data

The amount of missing data during the primary efficacy analysis period is expected to be very low due to the protocol-required 72-hour hospitalization of all subjects following surgery.

For any data that is missing through 72 hours in subjects who complete the 72-hour postoperative observation period, the NRS-R pain intensity scores will be imputed via last observation carried forward (LOCF), in which the most recent postdose nonmissing value is used for a subsequent missing value. If there is no postdose value available prior to the first missing value, then the median of values from subjects with observed values within the same treatment group at the relevant timepoint will be used. Predose values will not be carried forward to postdose timepoints.

In subjects who withdraw from the study prior to 72 hours, missing NRS-R pain intensity scores through 72 hours that were to be collected following withdrawal will be imputed via worst observation carried forward (WOCF), in which the worst (highest) NRS-R pain intensity score observed prior to withdrawal will be used for post-withdrawal values through 72 hours. Any missing NRS-R pain intensity scores prior to the point of withdrawal will be imputed via LOCF.

A table displaying the number and percentage of subjects with missing NRS-R pain intensity scores at each nominal timepoint will be produced.

All safety results will be summarized using observed cases with no imputation.

For partial dates involving AE start dates and concomitant medication start dates, the algorithms for imputation will vary depending upon the parameter; the details can be found in Appendix 1. No other partial dates will be imputed.

#### 6. SUBJECT DISPOSITION

A summary of disposition of subjects will include the number and percentage of subjects for the following categories: subjects enrolled (signed the Informed Consent Form), subjects who failed screening with reasons for screen failure, subjects in the Safety Population, subjects completing the 72-hour postoperative observation period, subjects completing Day 28, and subjects not completing Day 28 by reason for withdrawal. Only 1 reason for study withdrawal will be recorded for each subject.

# 7. DEMOGRAPHICS, CHARACTERISTICS, AND MEDICAL HISTORY

## 7.1. Demographics and Baseline Characteristics

Demographics and baseline characteristics will be presented in tables using descriptive statistics. Demographics consist of age, age category, sex, race, and ethnicity. Baseline characteristics consist of weight, height, and body mass index (BMI). A subject's age in years is calculated using the integer part of the difference in number of days between the date that informed consent is signed and date of birth divided by 365.25, or is recorded directly on the eCRF. The number and percentage of subjects in the following age categories will be presented: 18-44, 45-54, 55-64, 65-74, 75-84, and ≥ 85.

## 7.2. Medical History

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®) version 19.1. Medical history will be summarized for the Safety Population and will display the number and percentage of subjects with a past and/or concomitant disease or past surgeries by System Organ Class (SOC) and preferred term (PT).

#### 7.3. Protocol Deviations

Deviations and violations from the protocol will be recorded. Protocol deviations will be classified into, but not necessarily limited to, the following categories:

- ICF procedures.
- Eligibility criteria.
- Prohibited concomitant medication/therapy.
- Laboratory assessment.
- Study procedure (eg, efficacy ratings).
- Safety reporting.
- Randomization/blinding
- Study drug dosing/administration
- Visit schedule/windows

Protocol deviations will be presented in a summary table by protocol deviation category.

#### 8. TREATMENTS AND MEDICATIONS

#### **8.1.** Prior and Concomitant Medications

Prior medications are defined as medications with a stop date occurring before Day 1. Concomitant medications are defined as medications that are ongoing on Day 1 or with a start date occurring on or after Day 1. Medications with start and stop dates which bracket

Day 1, or for which missing start and/or stop dates make it impossible to determine the prior or concomitant status, will be summarized as concomitant medications.

All medications will be coded with the World Health Organization Drug Dictionary Enhanced (WHODDE), September 1, 2016.

Prior and concomitant medications will be summarized separately by drug class and PT. At each level of summarization, a subject is counted once if that subject reports 1 or more medications at that level. Drug class will correspond to the Anatomical Therapeutic Classification (ATC) Level 2 term.

Average daily use and total use of protocol-specified postoperative analysis medication will also be summarized using descriptive statistics for each analysis (ibuprofen and acetaminophen) for hours 0-24, 0-48, and 0-72.

## 8.2. Surgery Procedure

The side of the body subject to the surgical procedure (left or right), type of mesh, and the duration of surgery will be summarized. Duration will be calculated as completion time minus start time, reported in minutes. In addition, summary statistics will be provided for length of incision in centimeters.

## 8.3. Study Drug

For all subjects, treatment will consist of a single dose of study drug. As such, extent of exposure will be reported in the CSR as the number of subjects who received the study drug in the Safety Population. A summary of treatment compliance will not be produced, as by definition it will be 100% for the Safety Population.

#### 9. EFFICACY ANALYSIS

All efficacy summaries will be performed on the Safety Population and summarized within cohort and overall if optional Cohorts 2 or 3 are activated.

All efficacy analyses will consist of reporting summary statistics in tables and figures.

## 9.1. Primary Efficacy Endpoint

The primary efficacy endpoint is the proportion of subjects receiving no opioid rescue from 0-72 hours.

#### 9.1.1. Primary Analysis

The following steps will be implemented to identify opioid rescue medication during 0-72 hours:

- 1. Select concomitant medications that are coded as an opioid analysis.
- 2. Identify rescue medications from Step 1 in which the start date/time of medication is within the 72-hour postoperative observation period (see Section 5.4.5 for details).

The proportion of subjects receiving no opioid rescue medication from 0-72 hours will be summarized.

## 9.2. Secondary Efficacy Endpoints

The secondary efficacy endpoints are:

- Total postoperative opioid consumption (in IV morphine equivalents [IV MME]) through 72 hours.
- Proportion of subjects receiving no opioid rescue over the following time intervals: 0-24 hours, 24-48 hours, 0-48 hours, 24-72 hours, 48-72 hours.
- Proportion of subjects receiving no opioid rescue from 0-72 hours who receive no opioid rescue through Day 10, and through Day 28.
- Proportion of subjects in severe pain (NRS-R ≥ 7) at any point in the first 72 hours postoperatively.

#### Total postoperative opioid consumption (in morphine equivalents) through 72 hours

Determination of morphine equivalents

Use of rescue medications will be summarized by preferred term. All opioid dosages and formulations will have the IV MME calculated (Opioid Morphine Equivalent Conversion Factors, Centers for Disease Control and Prevention, Atlanta, GA, May 2014).

Table 1 displays the IV MME of selected opioid rescue medications. Protocol-allowed postoperative opioid rescue medications are checked. Opioid medications that are not protocol-allowed will be logged as protocol deviations, but will still be subject to IV MME conversion for analysis.

Table 1. Analgesic Windows and IV Morphine Milligram Equivalents for Opioid Rescue Medications in Preferred Terms

| Medication | Route | IV MME Factor | <b>Protocol Allowed</b> |
|---|---|---|---|
| CODEINE | PO | 0.05 | |
| HYDROMORPHONE HYDROCHLORIDE | PO | 1.33 | |
| HYDROMORPHONE HYDROCHLORIDE | IV | 6.67 | |
| FENTANYL | IV | 50.00 | |
| HYDROCODONE | PO | 0.40 | |
| MORPHINE | IV | 1.00 | ✓ |
| MORPHINE | PO | 0.33 | |
| MORPHINE | IM | 1.00 | |
| MORPHINE | PR | 1.00 | |
| OXYCODONE | IV | 1.00 | |
| OXYCODONE | IM | 1.00 | |
| OXYCODONE | PO | 0.50 | ✓ |
| PETHIDINE | IV | 0.13 | |
| TRAMADOL | IV | 0.06 | |
| TRAMADOL | РО | 0.04 | |

Protocol-allowed postoperative rescue medications consist of oral (PO) immediate-release oxycodone (no more than 10 mg within a 4-hour period as needed) or IV morphine (no more than 10 mg within a 2-hour period as needed). Administration of other opioids or any other analgesics (eg, ketamine, pregabalin), local anesthetics, or anti-inflammatory agents (except as specified by the protocol) is prohibited, unless needed to treat an AE that occurs after signing the ICF, for pretreatment prior to a needle placement, or to decrease venous irritation (eg, caused by propofol, in which case no more than a single administration of lidocaine 1% 20 mg IV may be administered). Combination opioid/non-opioid products (eg, Percocet) are not allowed.

#### Analysis method

Average daily use and total use of opioid rescue medication will be tabulated using descriptive statistics for each opioid and for overall opioids during the following periods: hours 0-24, hours 24-48, hours 0-48, hours 24-72, hours 48-72, and hours 0-72. Subjects who did not use a specific rescue medication during a period of interest will have their dose set to 0 for that period.

The mean total postoperative opioid consumption will also be plotted in a bar chart for hours 0-24, hours 0-48 and hours 0-72 with associated SEs.

# Proportion of subjects receiving no opioid rescue medication over the following time intervals: 0-24 hours, 24-48 hours, 0-48 hours, 24-72 hours, 48-72 hours

The proportion of subjects receiving no opioid rescue medication over these time periods will be summarized. The proportions of subjects receiving no opioid rescue medication from 0-24, 0-48, and 0-72 hours will be plotted in a bar chart. In addition, the proportions of subjects receiving no opioids from Day 1-10 and from Day 1-28 will be summarized. The Day 10 and Day 28 opioid use data will come from the subject diary.

# Proportion of subjects receiving no opioid rescue medication from 0-72 hours who receive no opioid rescue through Day 10, and through Day 28

Using the number of subjects receiving no opioid rescue medication from 0-72 hours as the denominator, the proportion of these subjects receiving no opioid rescue medication through Day 10 and through Day 28 will be summarized.

# Proportion of subjects in severe pain (NRS-R $\geq$ 7) at any point in the first 72 hours postoperatively

Acute severe pain at rest will be assessed through 72 hours following surgery. Proportions of subjects with an NRS-R score  $\geq$  7 at any time during hours 0-24, 0-48, and 0-72 will be summarized and plotted in a bar chart. In addition, a line plot of NRS-R pain intensity scores from hours 0-72 will be produced.

#### 10. SAFETY ANALYSIS

All analyses of safety data will be conducted using the Safety Population. No imputation of missing safety data will be performed except in the case of partial AE and concomitant medication onset dates (Appendix 1).

#### 10.1. Adverse Events

An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A TEAE is any AE which occurs any time during or after study drug administration, or any AE with an onset prior to study drug administration that worsens during or after study drug administration. An AE may be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not considered causally associated with the use of the study drug. Any abnormal laboratory value, or vital sign result deemed clinically significant by the Investigator, regardless of causal relationship, must be reported as an AE.

For an event to be a TEAE, it must meet one of the following conditions:

- Begins on Study Day 1, during or after administration of study drug.
- Begins after Study Day 1.
- Begins before Study Day 1 and worsens in severity during or after the Study Day 1 administration of study drug.

AEs with unknown onset dates or unknown end dates will be counted as TEAEs unless the event resolves before Study Day 1.

AEs will be coded using MedDRA version 19.1. Only TEAEs will be presented in AE tables, according to the SOC and PT. Any AEs that occur and resolve prior to Study Day 1 or are ongoing but do not worsen on or after Study Day 1 will be considered pretreatment AEs and will appear in the AE listing but not in TEAE tables.

#### **10.1.1.** Incidence of Treatment Emergent Adverse Events

The incidence of TEAEs table will include only 1 occurrence of a PT per subject. If a subject reports the same PT multiple times, then that PT will only be incremented by 1 since subject counts will be presented. As with the PT, if a subject reports multiple TEAEs within the same SOC, then that SOC will only be incremented by 1 since subject counts will be presented. For tables showing incidence by SOC and PT, SOCs will be sorted by the internationally agreed order and PTs will be sorted within SOC in descending order of incidence. For tables showing incidence by PT only, the PTs will be sorted in descending order of incidence.

An overall summary of TEAEs will be presented, and will include the following:

- Number of TEAEs.
- Number of subjects with at least 1 TEAE.
- Number of subjects with at least 1 possibly related TEAE.
- Number of subjects with at least 1 severe TEAE.
- Number of subjects with at least 1 TEAE leading to study withdrawal.
- Number of subjects with at least 1 ORAE.
- Number of subjects with at least 1 local inflammatory TEAE.
- Number of subjects with at least 1 potential LAST-related TEAE.
- Number of SAEs.
- Number of subjects with at least 1 SAE.
- Number of subjects with at least 1 possibly related SAE.
- Number of subjects with fatal TEAEs.

The incidence of all TEAEs will be presented by SOC and PT and separately by PT only.

#### 10.1.2. Relationship of Adverse Events to Investigational Drug

The incidence of possibly related TEAEs will be presented in a table by SOC and PT. TEAEs that are missing relationship will be considered "Possibly Related" for the purpose of this incidence table but will be presented in the data listing with a missing relationship.

#### **10.1.3.** Severity of Adverse Event

The incidence of severe TEAEs will be presented in a table by SOC and PT. TEAEs that are missing severity will be considered "severe" for the purpose of this incidence table but will be presented in the data listing with a missing severity.

#### 10.1.4. Serious Adverse Events

The seriousness of a TEAE should be assessed by the Investigator independently from the severity of the TEAE. An SAE is an AE occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing inpatient hospitalization, results in persistent or significant disability/incapacity, or is a congenital abnormality/birth defect.

Important medical events that may not be immediately life-threatening or result in death, or require hospitalization may be considered SAEs when, based upon medical judgment, they may jeopardize the subject or may require intervention to prevent one of the outcomes listed above.

SAEs will be presented in a listing.

#### **10.1.5.** Adverse Events Leading to Study Withdrawal

All TEAEs reported with "Withdrawal from Study" checked on the eCRF will be presented in a listing.

#### 10.1.6. Opioid-related Adverse Events

Incidence of TEAEs that are potentially opioid-related, regardless of whether a subject actually received an opioid medication, will be presented by PT. Prespecified PTs that may be opioid-related include the following:

- Nausea
- Vomiting
- Constipation
- Pruritus
- Pruritus generalised
- Somnolence
- Respiratory depression
- Urinary retention

Incidence of ORAEs will be presented separately as follows:

- Incidence of ORAEs.
- Incidence of ORAEs through the 72-hour postoperative observation period.

### **10.1.7.** Local Inflammatory Adverse Events

To enable a broad and comprehensive analysis of TEAEs potentially related to adverse effects on wound healing, local inflammatory TEAEs will be reviewed by searching the clinical database using a custom list of PTs created by Heron (Table 2).

Table 2. Local Inflammatory Adverse Events by Preferred Term

| <ul><li>Blister</li><li>Blood blister</li></ul> | Incision site haemorrhage Incision site infection | Postoperative wound infection |
|---|---|---|
| Cellulitis | Incision site oedema | Post procedural cellulitis |
| • Erythema <sup>a</sup> | Incision site rash | Purulent discharge |
| Impaired healing | Incision site swelling | Wound complication |
| Incision site cellulitis | Incision site vesicles | Wound dehiscence |
| Incision site | Infection | Wound infection |
| complication | Postoperative wound | Wound secretion |
| • Incision site erythema | complication | |

<sup>&</sup>lt;sup>a</sup> The Preferred Term of erythema was included in addition to incision site erythema for the most comprehensive review.

Incidence of local inflammatory TEAEs will be presented in a table by SOC and PT.

#### 10.1.8. Potential Local Anesthetic Systemic Toxicity (LAST) related Adverse Events

The symptoms that are potentially related to LAST will be reviewed by searching the clinical database using a custom list of PTs created by Heron (Table 3).

Table 3. Potential LAST-Related Adverse Events by Preferred Term

| • | Arrhythmia (any preferred term | • | Hypotension | • | Seizure |
|---|---|---|---|---|---|
| | with the string of "Arrhythmia") | • | Muscle twitching | • | Tinnitus |
| • | Bradycardia (any preferred term with the string of "Bradycardia") | • | Paraesthesia | • | Tremor |
| | • • • | • | Paraesthesia oral | • | Vision blurred |
| • | Cardiac arrest | | Respiratory arrest | | Visual impairment |
| • | Dizziness | | Respiratory arrest | | v isaar impairment |
| • | Dysgeusia | | | | |

Incidence of potential LAST-related TEAEs will be presented in a table by SOC and PT.

#### 10.1.9. Death

Any subject deaths during this study will be collected and presented in a listing. The information that is presented will include date of death, days on study, cause of death (AE preferred term), and relationship of death to study drug.

### 10.2. Clinical Laboratory Evaluations

Laboratory assessments will be performed by a central laboratory (hematology and serum chemistry) or locally (pregnancy test and drug screen). All summaries of central laboratory data will be based on the standard international (SI) units provided by the central lab. Associated laboratory parameters such as hepatic profile, renal function, and hematology values will be grouped and presented together.

Summary tables for hematology and chemistry including actual values and change from Baseline values will be presented for clinical laboratory tests with numeric values. These tables will include each visit (Baseline, Hour 72, and Day 10), highest postdose value, lowest postdose value, and last postdose value. Hematology will additionally include Hour 24.

Laboratory data will also be summarized using shift tables where appropriate. Each subject's hematology and serum chemistry values will be flagged as "low", "normal", or "high" relative to the normal ranges of the central laboratory.

Laboratory data collected at unscheduled visits will be included in listings and will contribute to tables of shifts from Baseline and in tables showing changes from Baseline to highest value, lowest value, and last value. Unscheduled laboratory results will not be windowed for the purposes of assigning a nominal visit.

Listings of laboratory values will include flags for values outside the central laboratory normal ranges that indicate how far out of the normal range an abnormal value is. For example, a value that is  $\geq 3$  times the upper limit of normal (ULN) but below 4 times the upper limit of normal will have a "3H" flag. Flag multipliers will show values that are 1, 2, 3, 4, 5, and 10 times relative to the ULN if high. Values that are below the lower limit of normal (LLN) will be flagged simply with "L".

Listings of abnormal values for hematology and chemistry will be presented separately in addition to listings of all laboratory values.

## 10.3. Hematology

The following laboratory tests will be included in hematology summary tables: hematocrit, hemoglobin, mean corpuscular volume (MCV), platelet count, red blood cell (RBC) count, and total and differential white blood cell (WBC) count (basophils, eosinophils, lymphocytes, monocytes, and neutrophils).

#### 10.3.1. Blood Chemistry

The following laboratory tests will be included in the blood chemistry summary tables: alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), bicarbonate, blood urea nitrogen (BUN), calcium, chloride, creatinine, direct bilirubin, gamma-glutamyltransferase (GGT), glucose, lactate dehydrogenase (LDH), magnesium, phosphorus, potassium, sodium, total bilirubin, total protein, and uric acid.

Associated laboratory parameters such as hepatic profile (ALT, albumin, ALP, AST, direct bilirubin, GGT, total bilirubin), electrolytes (bicarbonate, calcium, chloride, magnesium,

phosphorus, potassium, sodium), renal profile (BUN, creatinine), and other (glucose, LDH, total protein, uric acid) will be sorted/grouped together in table and listing presentations.

Evaluation of drug-induced serious hepatotoxicity (eDISH) scatterplots of the highest postdose ALT vs. total bilirubin observed at the same draw as the high ALT value, and of the highest postdose AST vs. total bilirubin observed at the same draw as the high AST value, will be produced.

The incidence of subjects with clinically relevant abnormalities in liver function tests will be summarized at each visit for the following categories. Subjects with clinical relevant abnormalities in Liver Function Tests will be presented in data listing as well.

- ALT or AST:
  - $\circ$  > 1 × ULN
  - $\circ \geq 2 \times ULN$
  - $\circ \geq 3 \times ULN$
  - $\circ \geq 4 \times ULN$
  - $\circ \geq 5 \times ULN$
- Total bilirubin  $\geq 2 \times ULN$
- ALP:
  - $\circ \geq 1.5 \times ULN$
  - $\circ \geq 2 \times ULN$
- ALT  $\geq$  3 × ULN and AST  $\geq$  3 × ULN
- ALT > 3 x ULN and total bilirubin  $> 2 \times ULN$
- AST  $\geq$  3 x ULN and total bilirubin  $\geq$  2 × ULN
- Potential Hy's Law: (ALT or AST  $\geq$  3 × ULN) and ALP < 2 × ULN and total bilirubin  $\geq$  2 × ULN

#### 10.3.2. Urine Pregnancy Test and Urine Drug Screen

Urine pregnancy test results (women of childbearing potential) and urine drug screen results will be listed.

#### 10.4. Vital Sign Measurements

Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate/pulse (HR), body temperature, and respiration rate will be collected at screening, on Day 1 before surgery, and post-treatment at 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 60, and 72 hours.

Summary tables including actual values and changes from Baseline will be presented for vital signs.

The number and percentage of subjects with clinically relevant abnormalities will be presented using data from any postdose visit (including unscheduled visits). Subjects with

clinical relevant abnormalities in vital signs will be presented in data listing as well. The criteria for clinically relevant abnormalities are shown in Table 4.

Table 4. Clinically Relevant Vital Signs Abnormalities

| Vital Sign | Low | High |
|---|---|---|
| HR | ≤50 bpm and ≥15 bpm decrease from Baseline | ≥120 bpm and ≥15 bpm increase from Baseline |
| SBP | ≤90 mmHg and ≥20 mmHg decrease from Baseline | ≥160 mmHg and ≥20 mmHg increase from Baseline |
| DBP | ≤50 mmHg and ≥15 mmHg decrease from Baseline | ≥100 mmHg and ≥15 mmHg increase from Baseline |

Abbreviations: bpm, beats per minute; DBP, diastolic blood pressure; HR, heart rate; SBP, systolic blood pressure.

## 10.5. Electrocardiogram

12-lead ECG (triplicate) is performed at screening and at 4, 24, 48, and 72 hours. ECG parameters include heart rate (beats/min), PR interval (ms), RR interval (ms), QRS interval (ms), QT interval (ms), and QTcF interval (ms). Overall interpretations of ECG results are also included.

ECG assessments will be performed in triplicate, and the mean value of the observed triplicates will be used for each ECG parameter. Summary statistics of ECG parameters and change from Baseline in ECG parameters will be presented using descriptive statistics at each scheduled visit. Shift from baseline of overall ECG interpretation at each postoperative timepoint will also be provided.

The number and percentage of subjects with clinically relevant abnormalities will be presented using summary table as well as data listing at each postoperative timepoint.

- QTcF values > 450 ms, > 480 ms, and > 500 ms
- Change from Baseline in QTcF values > 30 ms and > 60 ms
- QT values > 500 ms

## 10.6. Physical Examination

Physical examination is performed at Screening, 72 hours, and early termination. Physical examination data will be listed only.

## 10.7. Wound Healing Assessment

Wound healing assessment according to the Southampton Wound Scoring System (Bailey, Karran et al. 1992) is performed at 72 hours, on Day 10, and on Day 28. A summary of

wound healing assessment results will be produced, showing the number and percentage of subjects at each visit by grade with subgrade breakdown.

#### 11. INTERIM ANALYSIS

## 11.1. Interim Analysis

No formal interim analyses are planned.

#### 11.2. Data Safety Monitoring Board

An independent Data Safety Monitoring Board (DSMB) will not be involved with the conduct of this study. The Sponsor will review tables and listings of accumulating data approximately monthly to check enrollment, adherence to follow-up schedule, and ongoing safety results.

#### 12. REFERENCES

Bailey, I. S., S. E. Karran, K. Toyn, P. Brough, C. Ranaboldo and S. J. Karran (1992). "Community surveillance of complications after hernia surgery." <u>BMJ</u> **304**(6825): 469-471.

#### APPENDIX 1. IMPUTATION OF PARTIAL AND MISSING DATES

#### Incomplete Dates of Adverse Event start

All AE onset dates must be entered on the eCRF as complete dates. In the rare case that all or part of an AE onset date is missing but an AE resolution date is present and after study drug administration then the AE onset date will be imputed as follows:

| Year of onset | Month of onset | Day of onset | Onset date to be imputed as |
|---|---|---|---|
| Missing | Missing | Missing | Date of SDA |
| year = year of SDA | Missing | Nonmissing | Date of SDA |
| year = year of SDA | Missing | Missing | Set month and day to those of SDA |
| year < year of SDA | Missing | Nonmissing | set month to December |
| year < year of SDA | Missing | Missing | set month and day to December 31 |
| year > year of SDA | Missing | Nonmissing | set month to January |
| year > year of SDA | Missing | Missing | set month and day to January 1 |
| year = year of SDA | Month = month of SDA | Missing | Set day as day of SDA |
| year = year of SDA | Month < month of SDA | Missing | Set day as last day of onset month |
| year = year of SDA | Month > month of SDA | Missing | Set day as first day of onset month |
| year < year of SDA | Nonmissing | Missing | Set day as last day of onset month |
| year > year of SDA | Nonmissing | Missing | Set day as first day of onset month |

SDA = study drug administration.

If AE resolution date is present and prior to study drug administration, no need to impute incomplete AE start date, as the AE is not treatment emergent and the event should be in the medical history.

#### **Concomitant Medications**

- If year and month are present and day is missing then set day to first day of month for start date, and set day to last day of month for end date.
- If year and day are present and month is missing then set month to January for start date, and set month to December for end date.
- If year is present and month and day are missing then set month and day to January 1 for start date, and set month and day to December 31 for end date.
- Completely missing dates will not be imputed.

If start date is completely missing and end date is not prior to study drug administration, then the medication will be classified as concomitant; if the end date is missing, then the medication will be classified as ongoing. Medications for which the start and end dates are completely missing will be classified as concomitant.

## APPENDIX 2. DOCUMENT REVISION HISTORY

| Version | Date | Notes/Revisions |
|---|---|---|
| 1 | 18 October 2018 | Initial version, based on protocol version 1 (31 August 2018) |

## Signature Page for VV-TMF-36894 v1.0

| Reason for signing: Approved | Name:<br>Role: B<br>Date of signature: 19-Oct-2018 19:29:50 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: Role: C perations Date of signature: 19-Oct-2018 19:35:38 GMT+0000 |

Signature Page for VV-TMF-36894 v1.0